CLINICAL TRIAL: NCT06093737
Title: Reducing Disparities in Disaster-Related Mental Health Burden: Adaptation of a Multi-level Intervention to Build Community-based Response Capacity
Brief Title: Strengthening Community Mental Health
Acronym: COPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louisiana State University and A&M College (Other)
Collaborators: National Academies of Sciences, Engineering and Medicine (Unknown); University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Jennifer Lauren Scott, Associate Professor, Louisiana State University and A&M College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRBAM-21-139105
Record Dates: First submitted 2023-10-12; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Mental Health; Emotional Wellbeing; Anxiety; Depression; Stress; Coping; Perceived Stress; Perceived Social Support
Keywords: mental health; community-based participatory research; emotional wellbeing; perceived stress
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPE Intervention (Experimental): Is a three session brief group psychoeducational intervention. Session 1 is 4 hours, Session 2 and 3 are 1.5 hours. It is delivered in groups of 8-15 people with sessions spaced 1 month apart.
  Interventions: Behavioral: COPE: Communities Organizing for Power through Empathy
- House Meeting Control (Active Comparator): Is a 1.5 hour group meeting delivered in groups of 8-15 people spaced 1 month apart.
  Interventions: Behavioral: COPE: Communities Organizing for Power through Empathy

INTERVENTIONS:
Behavioral: COPE: Communities Organizing for Power through Empathy — A three session brief group psychoeducational intervention. Session 1 is 4 hours, Session 2 and 3 are 1.5 hours. It is delivered in groups of 8-15 people with sessions spaced 1 month apart.

SUMMARY:
The goal of this clinical trial is to examine the impact of the Communities Organizing for Power through Empathy (COPE) intervention in adults in communities having recently experienced or at risk of experiencing disaster. The main questions it aims to answer are:

* How does the COPE intervention affect individual mental health?
* How does the COPE intervention affect protective factors like coping and social support?
* How does the COPE intervention affect community resilience?
* How does delivery of the COPE intervention in partnership with a broad-based organization affect participant recruitment and retention, as well as outcomes?

Participants will participate in the three session COPE intervention. Researchers will compare individuals who participate in the COPE intervention to individuals who participate in house meetings to see if the COPE intervention improves mental health, coping, social support and community resilience. Researchers will also examine factors that affect implementation and intervention delivery.

DETAILED DESCRIPTION:
This Community-Based Participatory Research (CBPR) study will follow a multiphase mixed-methods design to adapt, deliver, and assess the efficacy of the Communities Organizing for Power through Empathy (COPE) intervention model. We will partner with a broad-based community organization, Together Baton Rouge, to adapt the intervention model to fit the context of East Baton Rouge Parish (EBRP) and deliver it to members of religious and non-profit institutions.

The objectives of the multi-level COPE intervention model are twofold: (1) reduce psychological distress and amplify protective factors among individuals and communities at risk of experiencing disasters; and (2) build individual and community psychological support response capacity. The intervention will be delivered by trained Community Facilitators (CFs) at community institutions (i.e., churches) to their institutional members. We will conduct a stepped wedge cluster randomized controlled trial (SWCRCT) to examine the impact of the COPE intervention. Measures of mental health, coping, social support and community resilience will be assessed at four timepoints (see timeline for data collection timepoints). We will conduct interviews and group reflections with CFs and participants to gain insight into their experiences with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years of age or older who are staff or members of an organization that is part of Together Baton Rouge and who participate in the intervention or are/were involved in the adaptation or implementation of the brief intervention in any capacity

Exclusion Criteria:

* Persons who are not 18 years of age or older and persons who are not staff or members of an organization that is part of Together Baton Rouge and/or not involved with the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in perceived stress from baseline | T1 (pre-intervention), T2 (1 month post-intervention), T3 (2 months post-intervention), T4 (3 months post-intervention)
  Measured using Perceived Stress Scale, a 10-item scale that measures the degree to which a person appraises situations in their life as stressful.
Change in depression symptoms from baseline | T1 (pre-intervention), T2 (1 month post-intervention), T3 (2 months post-intervention), T4 (3 months post-intervention)
  Measured using The Depression, Anxiety, and Stress Scale (DASS), a set of three self-report scales designed to measure depression, anxiety and stress.
Change in anxiety symptoms from baseline | T1 (pre-intervention), T2 (1 month post-intervention), T3 (2 months post-intervention), T4 (3 months post-intervention)
  Measured using The Depression, Anxiety, and Stress Scale (DASS), a set of three self-report scales designed to measure depression, anxiety and stress.
Change in stress symptoms from baseline | T1 (pre-intervention), T2 (1 month post-intervention), T3 (2 months post-intervention), T4 (3 months post-intervention)
  Measured using The Depression, Anxiety, and Stress Scale (DASS), a set of three self-report scales designed to measure depression, anxiety and stress.
Change in perceived social support from baseline | T1 (pre-intervention), T2 (1 month post-intervention), T3 (2 months post-intervention), T4 (3 months post-intervention)
  Measured using the Multidimensional Scale of Perceived Social Support (MSPSS) is a 12 item scale, assessing perceived social support and connection.
Change in coping from baseline | T1 (pre-intervention), T2 (1 month post-intervention), T3 (2 months post-intervention), T4 (3 months post-intervention)
  Measured using the Coping Self-Efficacy Scale (CSES) short form, a 12-item measure of confidence in managing stressors.
Change in community resilience from baseline | T1 (pre-intervention), T2 (1 month post-intervention), T3 (2 months post-intervention), T4 (3 months post-intervention)
  Measured using the Communities Advancing Resilience Toolkit (CART), a 21-item measure of community resilience items across 4 interrelated domains that both reflect and contribute to community resilience: (1) Connection and Caring; (2) Resources; (3) Transformative Potential; and (4) Disaster Management.

SECONDARY OUTCOMES:
Intervention acceptibility | After delivery of 3rd session
  Measured using the Acceptability of Intervention Measure (AIM), a 4 item measure of agreement with intervention.
Intervention appropriateness | After delivery of 3rd session
  Measured using the Appropriateness Measure (IAM), a 4 item measure of agreement with the appropriateness of the intervention.
Intervention feasibility | After delivery of 3rd session
  Measured using the Feasibility of Intervention Measure (FIM), a 4 item measure of agreement with the feasibility of implementing the intervention.

OTHER OUTCOMES:
Interviews | From date of first intervention delivery until 3 months post-date of delivery of final intervention session
  Semi-structured interviews about experience with participating in or facilitating the intervention
Focus groups | From date of first intervention delivery until 3 months post-date of delivery of final intervention session
  Periodic reflections conducted with community facilitators.
Intervention fidelity | At each intervention session.
  Assessed via facilitator observation using a structured fidelity questionnaire/form.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Scott, PhD, LCSW, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- Together Baton Rouge, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scott J, Powell T, Lee-Johnson NM. The Communities Organizing for Power Through Empathy (COPE) Community-Based Intervention to Improve Adult Mental Health During Disasters and Crises: Protocol for a Stepped-Wedge Cluster Randomized Trial. JMIR Res Protoc. 2025 May 20;14:e63723. doi: 10.2196/63723. PMID 40392582